CLINICAL TRIAL: NCT03524599
Title: Scale-up of Prevention and Management of Alcohol Use Disorders and Comorbid Depression in Latin America
Acronym: SCALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Newcastle University (Other); Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMFHMLCapH2020
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
Keywords: Heavy drinking; Primary health care; Training; Community
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention municipality (Experimental): In the intervention municipalities, primary health care providers will receive ongoing training and support in undertaking screening and brief advice for heavy drinking. They will also receive community-based five adoption mechanisms and five support systems.
  Interventions: Other: Intervention municipality
- Comparator municipality (No Intervention): In the comparator municipalities, the primary health care providers will be given a summary card of screening and brief advice for heavy drinking, with no instruction

INTERVENTIONS:
Other: Intervention municipality — In intervention municipalities, primary health care centres and the providers working within them will receive training and a range of community support mechanisms.
  Arms: Intervention municipality

SUMMARY:
A quasi-experimental study will compare primary health care-based prevention and management of alcohol use disorder, operationalized by heavy drinking, in three intervention cities from Colombia, Mexico and Peru with three comparator cities from the same countries. In the implementation cities, primary health care units (PHCUs) will receive training embedded within ongoing supportive municipal action over an 18-month implementation period. In the comparator cities, practice as usual will continue at both municipal and PHCU levels. The primary outcome will be the proportion of consulting adult patients intervened with (screened and advice given to screen positives).

ELIGIBILITY:
Inclusion Criteria:

* Any fully trained medical practitioner, nurse or practice assistant
* Non-temporary employment contract
* Working in the selected primary health care centre
* Involved in medical and/or preventive care

Exclusion Criteria:

* Not a fully trained medical practitioner, nurse or practice assistant
* Having a temporary employment contract
* Not working in the selected primary health care centre
* Not involved in medical and/or preventive care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of consulting adult patients (aged 18+ years) intervened | 18 months
  The number of AUDIT-C positive patients that received oral advice or referral for advice to another provider in or outside the primary health care centre (PHCC), divided by the total number of adult consultations of the participating providers per provider and per PHCC

SECONDARY OUTCOMES:
Proportion of patients screened | 18 months
  The proportion of patients screened will be calculated as the number of completed screens divided by the total number of consultations of all adult patients per participating provider, and averaged per participating PHCC
Proportion of patients advised | 18 months
  The proportion of patients advised will be calculated as the number of brief interventions delivered (received oral brief advice, and/or were referred to another provider in or outside the practice), divided by the total number of screen positives per participating provider and averaged per participating PHCC

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderson, MD, PhD, Principal Investigator — Professor
Locations (1):
- Health Services Unit Fray Bartolomé de las Casas, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solovei A, Jane-Llopis E, Mercken L, Bustamante I, Kokole D, Mejia-Trujillo J, Medina Aguilar PS, Natera Rey G, O'Donnell A, Piazza M, Schmidt CS, Anderson P, de Vries H. Effect of Community Support on the Implementation of Primary Health Care-Based Measurement of Alcohol Consumption. Prev Sci. 2022 Feb;23(2):224-236. doi: 10.1007/s11121-021-01329-1. Epub 2022 Jan 15. PMID 35032246
- [Derived] Anderson P, Manthey J, Llopis EJ, Rey GN, Bustamante IV, Piazza M, Aguilar PSM, Mejia-Trujillo J, Perez-Gomez A, Rowlands G, Lopez-Pelayo H, Mercken L, Kokole D, O'Donnell A, Solovei A, Kaner E, Schulte B, de Vries H, Schmidt C, Gual A, Rehm J. Impact of Training and Municipal Support on Primary Health Care-Based Measurement of Alcohol Consumption in Three Latin American Countries: 5-Month Outcome Results of the Quasi-experimental Randomized SCALA Trial. J Gen Intern Med. 2021 Sep;36(9):2663-2671. doi: 10.1007/s11606-020-06503-9. Epub 2021 Jan 19. PMID 33469752